CLINICAL TRIAL: NCT04837209
Title: A Phase II Study of NirAparib, Dostarlimab and Radiotherapy in Metastatic, PD-L1 Negative or Immunotherapy-Refractory Triple-Negative Breast Cancer (NADiR)
Brief Title: Radiation, Immunotherapy and PARP Inhibitor in Triple Negative Breast Cancer
Acronym: NADiR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Sibley Memorial Hospital (Unknown); Duke University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Steven J Isakoff, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-649
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — niraparib; dostarlimab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib + Dostarlimab + Radiation therapy (Experimental): Study cycle length is 3 weeks. Participants will receive:
  * Niraparib 1x daily during each study cycle
  * Dostarlimab 1x every 3 weeks for 4 study cycles, then 1x every 6 weeks beginning on Cycle 5
  * Radiation therapy will be given on Days 1, 2, and 3 of Cycle 1.
  Interventions: Drug: Niraparib; Drug: Dostarlimab; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Niraparib — Capsule, taken by mouth
  Other Names: Zejula
Drug: Dostarlimab — Intravenous infusion
  Other Names: TSR-042; WBP-285
Radiation: Radiation therapy — Radio Therapy

SUMMARY:
This research study is looking to see whether the combination of Dostarlimab and Niraparib plus Radiation Therapy (RT) is safe and effective in participants with metastatic triple negative breast cancer.

The names of the study treatment involved in this study are:

* Dostarlimab
* Niraparib
* Radiation Therapy (RT), which is given per standard of care.

DETAILED DESCRIPTION:
This is an open-label, phase II study that will evaluate how safe and well the combination of niraparib, dostarlimab, and Radiation Therapy (RT) works in metastatic triple negative breast cancer.

Niraparib is a type of drug called a "PARP inhibitor", which blocks DNA (the genetic material of cells) damage from being repaired or may prevent damage from occurring in the first place. In cancer treatment, inhibiting PARP may help kill cancer cells by not allowing the cancer cells to repair its DNA damage or prevent DNA damage associated with metastatic triple negative breast cancer from occurring.

Dostarlimab is a type of immunotherapy. It is believed to work by inhibiting (stopping) a protein called PD-1 from working. The PD-1 protein controls parts of the immune system (the system in a person's body that fights against diseases) by shutting down certain immune responses that are responsible for recognizing and destroying cancer cells.

The investigators believe that dostarlimab may inhibit the PD-1 protein on triple negative breast cancer cells, thus allowing the immune cells to recognize and destroy cancer cells.Radiation therapy is a standard-of-care treatment that is given to stop the growth of tumors. Radiation therapy can also stimulate the immune system, which leads to the destruction of tumor cells in the treated areas. Combining radiation therapy with anti-cancer drugs like dostarlimab and niraparib may increase the ability of the immune system to control or destroy cancer cells throughout the body.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive the study drugs for up to 2 years or until their triple negative breast cancer worsens Participants will then be followed for up to 5 years.

It is expected that about 32 people will take part in this research study.

The FDA has not approved niraparib for metastatic triple negative breast cancer, but it has been approved for other uses.

The U.S. Food and Drug Administration (FDA) has not approved dostarlimab as treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* ECOG performance status ≤ 1
* Histologically or cytologically-confirmed TNBC (ER <1%, PR <1%, HER-2-neu 0-1+ by IHC or non-FISH-amplified63. ER-low, PR-low (defined as ER and/or PR 1-10%) and HER2-negative patients may also be eligible, as per treating MD discretion).
* Metastatic or recurrent TNBC.
* Prior progression on immune-checkpoint inhibitor and/or PDL1-negative. Note: PDL1-status may be determined on tissues from either primary or mTNBC. PD-L1 status must be determined by an FDA-approved assay approved for breast cancer, such as PharmDx IHC (22C3) for pembrolizumab, Ventana (SP142) for atezolizumab
* No more than 2 prior lines of systemic therapy for inoperable/recurrent or metastatic disease.

Note: Prior line of systemic therapy includes targeted or biologic agents in combination or the absence of chemotherapy

* Radiation is clinically indicated for local control or palliation.
* At least one tumor for which RT is considered clinically appropriate.
* At least one radiographically-confirmed metastases index lesion that will not undergo RT and is measurable based on RECIST v1.1.
* Prior therapy with targeted agents or other forms of immunotherapy is allowed
* Prior RT is permitted, provided the treating radiation oncologist deems that study RT treatment planning guidelines can be achieved.
* Available archived tumor tissue of a metastatic tumor collected up to 28 days prior to registration. If archival tissue is unavailable, participant willingness to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 28 days prior to study registration.
* Adequate organ function (assessed within 8 days prior to initiation of protocol treatment, unless otherwise indicated) as follows:

  * Hematology

    * Absolute Neutrophil Count (ANC) ≥1500/mm3
    * Platelet Count ≥100,000/mm3
    * Hemoglobin ≥9.0 g/dL
  * Renal Function

    * Serum Creatinine ≤ 1.5 x upper limit of normal (ULN) or
    * Measured or calculated a creatinine clearance ≥ 60 mL/min for participant with (GFR can also be used in place of creatinine creatinine levels > 1.5 X ULN or CrCl
  * Hepatic Function

    * Total Bilirubin ≤ 1.5 mg/dL (Direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 ULN)
    * INR, PT, aPTT ≤ 1.5 x ULN (participants receiving anticoagulant therapy must have PT or PTT within therapeutic range)
    * Albumin ≥ 2.5 mg/dL
    * Aspartate Aminotransferase (AST) ≤ 2.5 x ULNb
    * Alanine Aminotransferase (ALT) ≤ 2.5 x ULNb ULN = upper normal limit of institution's normal range

      1. Creatinine clearance should be calculated per institutional standard.
      2. Participants with liver metastases may have AST and/or ALT ≤ 5 x ULN
* Female participant has a negative urine or serum pregnancy test within 7 days prior to study treatment if a woman has child-bearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment or is of non-childbearing potential.

Non-childbearing potential is defined as follows (by other than medical reasons):

* ≥45 years of age and has not had menses for >1 year
* Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.

  * Women of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 180 days after the last dose of study medication. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.

* Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 90 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Male subjects must not donate sperm starting with the first dose of study drug through 90 days after the last dose of study drug.
* Participant must agree not to breastfeed during the study or for 30 days after the last dose of study treatment.
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Ability to swallow (whole) and retain oral medications.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded:

* Known germline or somatic BRCA mutation-positive status
* Known active brain metastases or LMD (leptomeningeal disease). Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging [using the identical imaging modality for each assessment, either MRI or CT scan] for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and have not been using steroids for at least 7 days prior to study treatment.
* Known additional malignancy that progressed or required treatment in the last 2 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Prior treatment with either a PARP inhibitor or ICI is permitted, however, prior receipt of both therapies is excluded
* Receipt of >2 lines of chemo in the metastatic setting (including targeted or biologic agents in combination or the absence of chemotherapy)
* Hypersensitivity to niraparib or dostarlimab components or its excipients.
* Participation in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks (or at least 5 half-lives from previous therapy) of the first dose of study treatment.
* Receipt of prior cytotoxic therapy or targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., > Grade 1 or at baseline) from adverse events due to a previously administered agent, including grade 2 alopecia.

Note: Participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

* Patients who have undergone any major surgery within 3 weeks prior to study entry: patients must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Use of local corticosteroid injections (e.g. intra-articular injections), inhaled, intranasal, ophthalmic, and topical corticosteroids, and subjects requiring corticosteroid pre-medication for hypersensitivity reactions (e.g. CT scan pre-medication) are allowed.
* Known history of/active, non-infectious pneumonitis requiring treatment with steroids or has history of/active interstitial lung disease.
* Active infection requiring systemic therapy.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Participant has a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression.

Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 180 days after the last dose of trial treatment.

* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HbsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Known history of active TB (Bacillus Tuberculosis)
* Receipt of a live vaccine within 14 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
* Participant must not have received colony stimulating factors (eg, granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
* Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Patient experienced ≥ Grade 3 immune-related AE with prior immunotherapy, with the exception of non-clinically significant lab abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR)-RECIST | Enrollment to end of treatment up to 5 years
  Primary endpoint of the study is ORR as measured by RECIST v1.1. ORR will be estimated with the 95% confidence interval, based on the exact binomial distribution

SECONDARY OUTCOMES:
Overall response rate (ORR) by irRECIST criteria | Enrollment to end of treatment up to 5 years
  Assessed by irRECIST (Immune-related Response Evaluation Criteria in Solid Tumors)
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | Enrollment to end of treatment up to 5 years
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting
Overall survival (OS) | First day of study treatment to the date of death due to any cause, assessed up to 5 years
  The OS rate will be estimated by the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation
Progression-free survival (PFS) | First day of study treatment to the date of disease progression or death due to any cause, whichever came first, assessed up to 5 years
  The PFS rate will be estimated by the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation

OTHER OUTCOMES:
Changes in TILs | Enrollment to end of treatment up to 5 years
  Evaluate CD8+/CD3+ T cell infiltration pre-treatment will be compared to CD8+/CD3+ T cell infiltration during treatment (week 7), and correlation with objective response
ctDNA | Enrollment to end of treatment up to 2 years
  To evaluate changes in ctDNA using a patient-specific NGS ctDNA assay

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Isakoff, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation